CLINICAL TRIAL: NCT06432673
Title: The Attractive 2 Trial - An Open-label, Randomised, 2-period Cross-over Trial to Assess the Pharmacokinetics of ATR-258 Oral Capsule vs. Oral Solution Formulations in Healthy Volunteers
Brief Title: The Attractive 2 Trial - Pharmacokinetics of ATR-258 Oral Capsule vs. Oral Solution Formulations in Healthy Volunteers
Acronym: Attractive 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atrogi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ATR-258-trial-2; 2023-508797-28-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-07; First posted 2024-05-29 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-05

CONDITIONS: Type2diabetes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants receive a single dose of ATR-28 in the order Oral capsule - Oral solution with a washout period in between.
  Interventions: Drug: ATR-258 Oral solution; Drug: ATR-258 Oral capsule
- Arm 2 (Experimental): Participants receive a single dose of ATR-28 in the order Oral solution - Oral capsule with a washout period in between.
  Interventions: Drug: ATR-258 Oral solution; Drug: ATR-258 Oral capsule

INTERVENTIONS:
Drug: ATR-258 Oral solution — Oral solution
Drug: ATR-258 Oral capsule — Oral capsule

SUMMARY:
This is a single-centre, open-label, randomised, 2-period cross-over, Phase 1 comparative trial to assess the ATR-258 pharmacokinetic (PK) parameters of an oral capsule formulation in comparison with an oral solution formulation, both given as single doses to healthy volunteers. The order of treatment, i.e., the treatment sequence capsule - solution or solution - capsule, will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Body mass index ≥ 18.5 and ≤ 30.0
* Medically healthy participant
* Willing to use of double barrier contraceptive method if of childbearing potential

Exclusion Criteria:

* History or clinical manifestation of any clinically significant disease
* History of dysphagia or any other swallowing disorder
* Current smokers or users of nicotine products
* History or manifestation of drug abuse, alcohol abuse and/or excessive intake of alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 48 hours
Peak Plasma Concentration (Cmax) | 48 hours

SECONDARY OUTCOMES:
Time to maximum plasma concentration (Tmax) | 48 hours
  Tmax
Half life in plasma (T1/2) | 48 hours
Apparent total body clearance following extravascular administration (CL/F) | 48 hours
Volume of distribution following extravascular administration (Vz/F) | 48 hours
Adverse events | 7 days post last dose
  Frequency, intensity and seriousness of reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Erik Waara, Study Chair — Atrogi AB
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No